CLINICAL TRIAL: NCT03185338
Title: A School-based Physical Activity Promotion Intervention in Children: Rationale and Study Protocol for the PREVIENE Project
Brief Title: A School-based Physical Activity Promotion Intervention in Children. PREVIENE Project
Acronym: PREVIENE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Pablo Tercedor, Professor, Universidad de Granada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEP2015-63988-R
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Motor Activity
Keywords: physical activity, promotion, school
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Active commuting to/from school (Experimental): This intervention will be focused on children and their families following the ecological model proposed by Sallis et al., targeting mainly individual factors such as children's perceptions (safety perception on the way to school) and attitudes (independence or motivation to walk). A total of six 1-hour activities will be conducted at the classroom and two activities in the school neighborhood designed based on previous literature. Taken together, these activities will emphasize the benefits of active commuting to/from school and promote active commuting to/from school.Moreover, supporting information will be sent to families on four occasions during the intervention to encourage families to use active modes of commuting to/from school.
  Interventions: Behavioral: Active commuting to/from school
- Active Physical Education lessons (Experimental): This intervention has been developed by the Spanish Ministry of Health, Social Services and Equality and the Ministry of Education, Culture and Sport to increase the amount of children's PA during PE lessons in primary schools. At the time of this study, any school in Spain could choose to adopt this programme. This intervention includes two sets of eight active PE lessons specifically developed for third grade of primary school. These lessons will replace the original PE lessons in schools assigned to Active PE lesson intervention and integrated intervention.Additionally, this intervention provides some methodological advices to increase the PA time during the PE lesson (i.e. different ways to take attendance or deciding on the most suitable activity given the availability of resources).
  Interventions: Behavioral: Active Physical Education lessons
- Active school recess (Experimental): This intervention has been designed based on previous research. The teacher will prepare the school playground offering adequate space and games to encourage children to be active. A sheet placed on the wall as a reminder will help teacher to remind children to participate and motivate them. On this sheet, each child will write the activity completed during the school recess every day during the intervention period.
  Interventions: Behavioral: Active school recess
- Sleep health promotion (Experimental): Eight activities will be carried out at home and at school. During the first activity, parents and children will attend a general talk about sleep and health and will sign a contract for a "healthy sleep at home". Also, children will complete a diary in which they will keep a record of their activities prior to going to bed and after waking up in the morning. At school, the first classroom-based activity will be based on the educational program "I have a dream" (Spanish adaptation of the SimplyHealthy@Schools International Program). The remaining classroom-based activities will include with a group art project with questions and answers about sleep, discussion groups about the sleep diary completed at home, and an abbreviated version of the Jacobson's progressive relaxation technique.
  Interventions: Behavioral: Sleep health promotion
- School global intervention (Experimental): Also, a simultaneous implementation of all four interventions (see the others arms) will be examined in one of the intervention schools.
  Interventions: Behavioral: Active commuting to/from school; Behavioral: Active Physical Education lessons; Behavioral: Active school recess; Behavioral: Sleep health promotion; Behavioral: School global intervention
- Control school (No Intervention): Control school will be evaluate but will not receive any intervention

INTERVENTIONS:
Behavioral: Active commuting to/from school — Active transport to/from school on foot or by bike will be promoted
  Arms: Active commuting to/from school; School global intervention
Behavioral: Active Physical Education lessons — Specific lessons designed for increasing moderate to vigorous physical activity in Physical Education will be applied
  Arms: Active Physical Education lessons; School global intervention
Behavioral: Active school recess — Teachers will design games and activities and will encourage children for being active
  Arms: Active school recess; School global intervention
Behavioral: Sleep health promotion — This intervention will aim to raise the awareness of the importance of having a good quality sleep at night and to teach healthy sleep behaviours that will contribute to improving sleep hygiene
  Arms: School global intervention; Sleep health promotion
Behavioral: School global intervention — A simultaneous implementation of all four interventions (see the others arms) will be examined in one of the intervention schools.
  Arms: School global intervention

SUMMARY:
Background:The lack of physical activity and increasing time spent in sedentary behaviours during childhood place importance on developing low cost,easy-to-implement school-based interventions to increase physical activity among children. The PREVIENE Project will evaluate the effectiveness of five innovative, simple, and feasible interventions(active commuting to school, Physical Education lessons, active school recess physical activity, sleep health promotion, and an integrated program incorporating all 4 interventions) to improve physical activity, fitness, anthropometry, sleep health, academic achievement,and health-related quality of life in primary school children.

Methods:A total of 350 children (grade 3; 8-9 years of age) from six schools in Granada (Spain) will be enrolled in one of the 8-week interventions (one intervention per school; 50 children per school) or a control group (no intervention school; 50 children). Outcomes will include physical activity (measured by accelerometry), physical fitness (assessed using the ALPHA fitness battery), anthropometry (height, weight and waist circumference), sleep health (measured by accelerometers, a sleep diary, and sleep health questionnaires), academic achievement (grades from the official school's records), and health-related quality of life (child and parental questionnaires).To assess the effectiveness of the different interventions on objectively measured PA and the other outcomes, the generalized linear model will be used.

Discussion: The PREVIENE Project will provide the information about the effectiveness and implementation of different school-based interventions for physical activity promotion in primary schoolchildren.

Keywords:children, physical activity, school,active commuting, Physical Education, school recess, sleep health, fitness, academic achievement, health-related quality of life.

DETAILED DESCRIPTION:
Background

The lack of physical activity and increasing time spent in sedentary behaviours during childhood place importance on developing low cost,easy-to-implement school-based interventions to increase physical activity among children. The PREVIENE Project will evaluate the effectiveness of five innovative, simple, and feasible interventions (active commuting to school, Physical Education lessons, active school recess physical activity, sleep health promotion, and an integrated program incorporating all 4 interventions) to improve physical activity, fitness, anthropometry, sleep health, academic achievement,and health-related quality of life in primary school children.

Methods

The PREVIENE Project uses a quasi-experimental approach with a convenience sample size of 300 children (grade 3, 8-9 years old) from six primary schools in Granada (Spain) (2 classes per school x 6 schools = 12classesin total). With the average class size of 25 children and the expected recruitment rate is 90%, two classes will be selected in each participating school. All 79 primary schools in Granada will be invited to participate in this study. The schools will initially be contacted by email followed by a phone call. Research team will arrange a meeting with the interested schools and their staff (principal, physical education teacher and other relevant teachers). At this meeting, the researchers will explain the main objective of this study and the inclusion criteria for schools' participation: 1) At least 2 classes of grade 3 children at school, 2) the average class size has to be 25 or more children. Once determined the schools that satisfy the inclusion criteria and express their willingness to participate, a total of six schools will be randomly selected.

The Regional Ministry of Education will endorse the participation of each selected school in the study. At the beginning of the study, families of all children in the selected classes will receive an invitation to an initial meeting at school to receive information about the study. Both children and parents will be encouraged to participate in the study. Parents will sign an informed consent which include the participation of them and their child. The study protocol has been approved by the University of Granada Human Research EthicsCommittee (Reference: 57/CEIH/2015).

Five schools will be randomly assigned to an intervention schools, four of them will apply a single intervention (n=50 children per intervention/school) and one school will implement the integrated program (all four interventions simultaneously;n=50 children).The sixth school will serve as a control school and will not receive any intervention (n=50 children). In schools assigned to the active PE lesson and integrated intervention, standard PE lessons will be replaced for the Active Didactics Unit. In all other schools, children will be exposed to the usual PE session's structure according to the National Education Program in Spain (i.e. 45 min sessions twice per week).

Interventions

Active commuting to/from school

This intervention will include a range of school-, family- and community-based activities. These activities will be focused on children and their families following the ecological model proposed by Sallis et al., targeting mainly individual factors such as children's perceptions (safety perception on the way to school) and attitudes (independence or motivation to walk). A total of six 1-hour activities will be conducted at the classroom and two activities in the school neighborhood designed based on previous literature. Taken together, these activities will emphasize the benefits of active commuting to/from school and promote active commuting to/from school using phrases such as "If you rides a bike for 1.200 km, the medium number of disease days will be reduced by one" for families.Moreover, supporting information will be sent to families on four occasions during the intervention to encourage families to use active modes of commuting to/from school. The supporting information will consist of sending messages by whatsapp and advices (text and images) explaining the most important ideas related active commuting and benefits of active commuting on academic achievements and children´s mental and physical health.

Finally, throughout the intervention period, the teacher will ask children their mode of transport to school of that day twice a week by raising their hand and encourage possible changes in mode of commuting as motivational strategy by using positive reinforcement (as reinforce when some children accompanied each other in the way to school). The objective of this reinforcement is to remind children to active commute to and from school.

Active PE lessons

This intervention has been developed by the Spanish Ministry of Health, Social Services and Equality and the Ministry of Education, Culture and Sport to increase the amount of children's PA during PE lessons in primary schools. At the time of this study, any school in Spain could choose to adopt this programme. This intervention includes two sets of eight active PE lessons specifically developed for third grade of primary school. These lessons will replace the original PE lessons in schools assigned to Active PE lesson intervention and integrated intervention. Additionally, this intervention provides some methodological advices to increase the PA time during the PE lesson (i.e. different ways to take attendance or deciding on the most suitable activity given the availability of resources).

Active school recess

This intervention has been designed based on previous research. The teacher will prepare the school playground offering adequate space and games to encourage children to be active. A sheet placed on the wall as a reminder will help teacher to remind children to participate and motivate them. On this sheet, each child will write the activity completed during the school recess every day during the intervention period.

Sleep health promotion

This intervention will aim to raise the awareness of the importance of having a good quality sleep at night and to teach healthy sleep behaviours that will contribute to improving sleep hygiene. As a part of this intervention, eight activities will be carried out at home and at school. During the first activity, parents and children will attend a general talk about sleep and health and will sign a contract for a "healthy sleep at home". Signing "the contract" will enable participants to have an active role in the sleep intervention. Also, with help of their parents at home, children will complete a diary in which they will keep a record of their activities prior to going to bed and after waking up in the morning. The objective of this activity is to strengthen the importance of a routine before going to sleep and its benefits on the adequate sleep behaviour. Parents will be given a manual to help children use an adequate sleep routine and reinforce children's achievements. At school, several teachers assisted by the researchers will implement the activities. The first classroom-based activity will be based on the educational program "I have a dream" (Spanish adaptation of the SimplyHealthy@Schools International Program; Philips Ibérica, S.A., Madrid, Spain). The remaining classroom-based activities will include with a group art project with questions and answers about sleep, children's calculation of their own sleep parameters from the sleep log data, and discussion groups about the sleep diary completed at home and other sleep issues, as well as strategies to achieve the commitments included in the "signed contract". In addition, the class teacher will introduce the concept of relaxation and its benefits at bedtime and will teach an abbreviated version of the Jacobson's progressive relaxation technique every morning after the recess.

School global intervention

Also, a simultaneous implementation of all four interventions (see the others arms) will be examined in one of the intervention schools.

Data analysis

Demographic characteristics will be analysed using descriptive statistics. Data will be presented using the mean and standard deviation or median and interquartile range, where appropriate for continuous variables, and frequency and percentage for categorical variables. To assess the effectiveness of the different interventions on objectively measured PA and the other outcomes, the generalized linear model will be used with the outcome measures as dependent variables in separate models, the intervention as an independent variable and controlling for potential confounders (such as gender, body mass index, socioeconomic status, and baseline PA). Statistical significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Schools with at least two groups of students
* Each group with at least 25 students

Exclusion Criteria:

* None

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2018-01-09 (Estimated); Primary Completion 2018-01-17 (Estimated); Study Completion 2019-10-22 (Estimated)

PRIMARY OUTCOMES:
Sedentary time | Change from baseline to week 8 and 5 months later
  Sedentary time will be measured using a tri-axial accelerometer (Actigraph wGT3X-BT, Pensacola, FL, USA) on 7 consecutive days, 24 hours/day. Children will be instructed to wear an accelerometer attached to the non-dominant wrist. Children will take it off only while water-based activities.Children will also complete a log to record the time when they take off the accelerometer. The results will be registered in minutes.
Light physical activity | Change from baseline to week 8 and 5 months later
  Light physical activity will be measured using a tri-axial accelerometer (Actigraph wGT3X-BT, Pensacola, FL, USA) on 7 consecutive days, 24 hours/day. Children will be instructed to wear an accelerometer attached to the non-dominant wrist. Children will take it off only while water-based activities.Children will also complete a log to record the time when they take off the accelerometer. The results will be registered in minutes.
Moderate physical activity | Change from baseline to week 8 and 5 months later
  Moderate physical activity will be measured using a tri-axial accelerometer (Actigraph wGT3X-BT, Pensacola, FL, USA) on 7 consecutive days, 24 hours/day. Children will be instructed to wear an accelerometer attached to the non-dominant wrist. Children will take it off only while water-based activities.Children will also complete a log to record the time when they take off the accelerometer. The results will be registered in minutes.
Vigorous physical activity | Change from baseline to week 8 and 5 months later
  Vigorous physical activity will be measured using a tri-axial accelerometer (Actigraph wGT3X-BT, Pensacola, FL, USA) on 7 consecutive days, 24 hours/day. Children will be instructed to wear an accelerometer attached to the non-dominant wrist. Children will take it off only while water-based activities.Children will also complete a log to record the time when they take off the accelerometer. The results will be registered in minutes.
Moderate-to-vigorous physical activity | Change from baseline to week 8 and 5 months later
  Moderate and vigorous physical activity will be combined to report moderate-to-vigorous physical activity

SECONDARY OUTCOMES:
Sociodemographic characteristics and health status | Change from baseline to week 8 and 5 months later
  Parents will complete a questionnaire about child's sociodemographic characteristics including date of birth and gender, household factors,family's socioeconomic characteristics (family income, parental education and parental employment status) and child's health status (reporting medical conditions and medications, if any).
Weight | Change from baseline to week 8 and 5 months later
  Weight will be assessed wearing PE clothes (shorts and a short sleeve shirt) and bare feet. Weight will be measured with a 0.1 kg approximation using a Seca 876 weighing system (Seca, Ltd., Hamburg, Germany).
Height | Change from baseline to week 8 and 5 months
  Height will be assessed wearing PE clothes (shorts and a short sleeve shirt) and bare feet. Height will be measured in the Frankfort plane, with an approximation of 0.1 cm using a Seca 2013 stadiometer (Seca, Ltd., Hamburg, Germany).
Body Mass Index | Change from baseline to week 8 and 5 months later
  Weight and height will be combined to report body mass index in kg/m^2
Waist circumference | Change from baseline to week 8 and 5 months
  Waist circumference will be assessed in a horizontal plane, at the level of the natural waist, by the measuring tape Seca 201 (Seca, Ltd., Hamburg, Germany)
Handgrip strength | Change from baseline to week 8 and 5 months later
  Handgrip strength will be assessed using the handgrip strength test included in ALPHA fitness test battery. The result will be registered in kilograms.
Explosive power of the legs | Change from baseline to week 8 and 5 months later
  Explosive power of the legs will be assessed using the standing long jump test included in ALPHA fitness test battery. The result will be registered in centimeters.
Speed-agility | Change from baseline to week 8 and 5 months later
  Speed-agility will be assessed using the 10-meter shuttle run test included in ALPHA fitness test battery. The result will be registered in centimeters.
Cardiorespiratory fitness | Change from baseline to week 8 and 5 months later
  Cardiorespiratory fitness will be assessed using the 20-meters shuttle run test included in ALPHA fitness test battery. The result will be registered in seconds.
Commuting to school behaviour | Change from baseline to week 8 and 5 months later
  Children will complete the questionnaire Pedalea y Anda al COlegio [ride a bike and go on foot to school] (PACO) with the help of the teacher and researcher at school. The Spanish and English versions of the questionnaire is available at http://profith.ugr.es/pages/investigacion/recursos/paco
Total sleep time | Change from baseline to week 8 and 5 months later
  Total sleep time will be assessed using accelerometry (ActigraphwGT3X-BT, Pensacola, FL, USA) 7 consecutive days, 24 hours/day. Children will be instructed to wear an accelerometer attached to the non-dominant wrist. The results will be registered in minutes.
Sleep onset latency | Change from baseline to week 8 and 5 months later
  Sleep onset latency will be assessed using accelerometry (ActigraphwGT3X-BT, Pensacola, FL, USA) 7 consecutive days, 24 hours/day. Children will be instructed to wear an accelerometer attached to the non-dominant wrist. The results will be registered in minutes.
Sleep efficiency | Change from baseline to week 8 and 5 months later
  Sleep efficiency will be assessed using accelerometry (ActigraphwGT3X-BT, Pensacola, FL, USA) 7 consecutive days, 24 hours/day. Children will be instructed to wear an accelerometer attached to the non-dominant wrist. The results will be registered in minutes.
Wake after sleep onset | Change from baseline to week 8 and 5 months later
  Wake after sleep onset will be assessed using accelerometry (ActigraphwGT3X-BT, Pensacola, FL, USA) 7 consecutive days, 24 hours/day. Children will be instructed to wear an accelerometer attached to the non-dominant wrist. The results will be registered in minutes.
Sleep knowledge and hygiene | Change from baseline to week 8 and 5 months later
  Children's sleep knowledge will be assessed using the Sleep Knowledge and Sleep Hygiene questionnaire developed by Philips as part of the educational program "I have a dream" (Spanish adaptation of the SimplyHealthy@Schools International Program; Philips Ibérica, S.A., Madrid, España). This questionnaire includes six questions about sleep knowledge and sleep-related behaviours (sleep hygiene, and bed time routine).
Pediatric Sleep Questionnaire | Change from baseline to week 8 and 5 months later
  Parents will complete the Pediatric Sleep Questionnaire to report general children's sleep behaviour, symptoms related to sleep disorders (especially, sleep apnea, enuresis, and parasomnias), and daytime behaviour hypersomnolence, inattention, hyperactivity). The questionnaire contains 71 items with response categories "yes", "no" and "don't know" and 18 four-point Likert-type items. This questionnaire has been validated in Spanish children
Pediatric Daytime Sleepiness Scale | Change from baseline to week 8 and 5 months later
  Parents will complete the Pediatric Daytime Sleepiness Scale to assesses daytime sleepiness-related behaviour. The scale contains 8 items answered by parents and scored from 0 to 4, using a 5-point Likert-scale. The questionnaire was translated into Spanish and has been tested for comprehension in Spanish children
Academic achievement | Change from baseline to week 8 and 5 months later
  Academic achievement will be determined from the final grades from the official school's records at the end of each trimester of the academic year in which data are collected. The academic indicators will be the grades (ranging from 0 to 10) from selected subjects (Natural Science, Social Sciences, Language (Spanish), Foreign language (English), Music, Arts and PE) and the medium grade (sum of the grade obtained in each of the subjects divided by the total of subjects).
Health-Related Quality of Life | Change from baseline to week 8 and 5 months later
  Health-related quality of life will be assessed using the Revidierter KINDer Lebensqualitätsfragebogen (KINDL-R), validated for 4 to 16 years old Spanish children.The KINDL-R consists of 24 items associated with 6 dimensions of health-related quality of life: physical well-being (e.g., illness, pain, fatigue), emotional well-being (e.g., boredom, loneliness, scared), self-esteem (e.g., pride, feeling on top of the world), family (e.g., relationship with parents, conflict at home), friends (e.g., getting along, feeling different from others), everyday functioning in school (e.g., enjoying class, worrying about the future) and disease (e.g., illness uncertainty, parent overprotection, missing school).Both children and parents will complete the respective versions of the KINDL-R questionnaires.The total score of both child and parental questionnaires will be transformed to a scale of 0 to 100, where higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tercedor, PhD, Principal Investigator — Universidad de Granada

IPD SHARING:
Plan to Share IPD: Undecided